CLINICAL TRIAL: NCT04980482
Title: A Randomized, Open-Label, Multicenter Study Investigating AB-729, Nucleos(t)Ide Analogue and Pegylated Interferon Alfa-2a Treatment in Subjects With Chronic Hepatitis B Infection
Brief Title: Open-Label Study of AB-729, Nucleos(t)Ide Analogue and Pegylated Interferon Alfa-2a in Subjects With Chronic Hepatitis B Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbutus Biopharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB-729-201
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Chronic Hepatitis b
Keywords: Hepatitis B virus; Chronic hepatitis B; HBV; Hepatitis; CHB
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort A, Group 1 (Experimental): AB-729 60 mg SC every 8 weeks + NA for 24 weeks, then randomized to:
  AB-729 60 mg SC every 8 weeks + NA + Peg-IFNα-2a 180 mcg SC every week for 24 weeks.
  Interventions: Drug: AB-729; Drug: Peg-IFNα-2a
- Cohort A, Group 2 (Experimental): AB-729 60 mg SC every 8 weeks + NA for 24 weeks, then randomized to:
  NA + Peg-IFNα-2a 180 mcg SC every week for 24 weeks.
  Interventions: Drug: AB-729; Drug: Peg-IFNα-2a
- Cohort B, Group 1 (Experimental): AB-729 60 mg SC every 8 weeks + NA for 24 weeks, then randomized to:
  AB-729 60 mg SC every 8 weeks + NA + Peg-IFNα-2a 180 mcg SC every week for 12 weeks.
  Interventions: Drug: AB-729; Drug: Peg-IFNα-2a
- Cohort B, Group 2 (Experimental): AB-729 60 mg SC every 8 weeks + NA for 24 weeks, then randomized to:
  NA + Peg-IFNα-2a 180 mcg SC every week for 12 weeks.
  Interventions: Drug: AB-729; Drug: Peg-IFNα-2a

INTERVENTIONS:
Drug: AB-729 — subcutaneous injection
Drug: Peg-IFNα-2a — subcutaneous injection
  Other Names: pegylated interferon alpha 2a

SUMMARY:
This is a randomized, open label, multicenter Phase 2 study investigating the safety and antiviral activity of AB-729 in combination with ongoing NA therapy and short courses of Peg-IFNα-2a in subjects with CHB.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B virus infection with documentation at least 6 months prior to screening
* Subjects must have been receiving either TAF, TDF (or equivalent), or ETV consistently for ≥12 months prior to dosing Day 1
* HBV DNA <LLOQ at Screening
* HBsAg between 100 and 5,000 IU/mL at Screening
* Subjects must be HBeAg-negative at Screening
* Fibroscan® result of ≤8.5 kPa within 6 months prior to dosing Day 1
* Medically stable based on physical examination, medical history, vital signs, laboratory values, and 12-lead Electrocardiogram (ECG) at screening

Exclusion Criteria:

* Evidence of co-infection with hepatitis A, C, D or E virus or human immunodeficiency virus (HIV) at screening
* History of any clinically significant medical condition associated with chronic liver disease, cirrhosis, evidence of decompensated liver disease, or findings suggestive of hepatocellular carcinoma (HCC) at any time
* Contraindications to the use of Peg-IFNα-2a or incapable of self-administration or assisted administration of Peg-IFNα-2a
* Previous treatment with an experimental HBV-directed RNA-interference or antisense oligonucleotide product.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
The frequency and severity of treatment emergent adverse events (TEAEs), discontinuations due to adverse events (AEs), and laboratory abnormalities after dosing with AB-729 plus Peg-IFNα-2a | Up to 124 weeks

SECONDARY OUTCOMES:
Change from baseline in HBsAg and other virologic markers at each time point | Up to 124 weeks
Proportion of subjects with HBsAb seroconversion at each timepoint | Up to 124 weeks
Proportion of subjects who are eligible to stop NA after Week 24 of follow up | Up to 76 weeks
Proportion of subjects who discontinue NA and subsequently restart NA therapy after meeting criteria | Up to 124 weeks
Proportion of subjects who discontinue NA and subsequently meet protocol defined clinical relapse criteria. Proportion of subjects who discontinue NA and subsequently meet protocol defined viral relapse criteria | Up to 124 weeks
Post-dose plasma concentrations of AB-729 anti-sense (AS), AB-729 AS(N-1)3', and AB-729 AS(N-2)3' at selected timepoints | Up to 40 weeks

CONTACTS AND LOCATIONS:
Locations (17):
- United States (6):
  - Arizona Liver Health, Chandler, Arizona
  - Arizona Liver Health, Tucson, Arizona
  - Research and Education, Inc., San Diego, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Henry Ford Health System, Detroit, Michigan
  - ID Care, Hillsborough, New Jersey
- Australia (2):
  - Nepean Hospital, Kingswood, New South Wales
  - St Vincent's Hospital Melbourne, Melbourne, Victoria
- Hong Kong (2):
  - Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Arensia Exploratory Medicine Moldova, Chisinau, Moldova
- South Korea (2):
  - Pusan National University Hospital, Pusan, Republic of Korea
  - Asan Medical Center, Seoul
- Taiwan (3):
  - Chia-Yi Christian Hospital, Chiayi City
  - Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
- Medical Center of Limited Liability Company Harmoniya Krasy, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No